CLINICAL TRIAL: NCT01139983
Title: Search for Novel Genes in Osteosarcoma Revealed by Analysis of Tumour Copy-Number Alterations and Constitutional Copy-Number Variations
Brief Title: DNA Biomarkers in Samples From Patients With Osteosarcoma and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST10B4; COG-AOST10B4 (Other: Children's Oncology Group); CDR0000674830 (Other: Clinical Trials.gov); NCI-2011-02234 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — In Situ Hybridization, Fluorescence; Microarray Analysis; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: fluorescence in situ hybridization
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying DNA biomarkers in samples from patients with osteosarcoma and healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether common copy-number alterations (CNAs) at chr7p14.1 arise de novo in osteosarcoma (OS) tumor DNA or whether they represent progression of constitutional copy-number variations (CNVs).
* To determine the association between constitutional CNVs at chr7p14.1 and susceptibility to OS.
* To determine how CNVs translate into CNAs in tumor DNA samples from patients with OS.

OUTLINE: RNA and DNA samples from banked blood and paired tumor tissue, plus samples from healthy controls, are analyzed for common copy-number alterations and constitutional copy-number variations (CNVs) at chr7p14.1 by microarray, q-PCR, RT-PCR, and FISH. Osteosarcoma predisposing CNVs results are then compared among cases versus healthy controls.

Clinical information associated with each osteosarcoma sample (i.e., gender, age of diagnosis, tumor site, tumor type and grade, presence of metastases at time of diagnosis, response to chemotherapy, event-free survival, and overall survival) is also collected, if available.

PROJECTED ACCRUAL: A total of 243 samples from patients with osteosarcoma and 80 samples from healthy controls will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of osteosarcoma (OS) and meets 1 of the following criteria:

    * Original 153 OS samples, including paired germline and tumor DNA
    * Additional samples from 90 patients with OS:

      * Blood samples
      * Germline DNA
      * Paired tumor biopsy tissue (not from resection) obtained before systemic chemotherapy
  * Healthy controls, age- and gender-matched

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-04; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Role of copy-number alterations (CNAs) in the etiology of osteosarcoma
Association between copy-number variations (CNVs) at chr7p14.1 and susceptibility to osteosarcoma
Relationship between CNVs and tumor CNAs in osteosarcoma

CONTACTS AND LOCATIONS:
Overall Officials: David Malkin, MD, Principal Investigator — The Hospital for Sick Children